CLINICAL TRIAL: NCT02908035
Title: TANGO: Temsirolimus Adventitial Delivery to Improve ANGiographic Outcomes Below the Knee
Brief Title: Temsirolimus Adventitial Delivery to Improve Angiographic Outcomes Below the Knee (TANGO)
Acronym: TANGO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mercator MedSystems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIP0214
Record Dates: First submitted 2016-09-16; First posted 2016-09-20 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Chronic Limb Ischemia
MeSH Terms: interventions — temsirolimus; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Active Comparator: Temsirolimus Delivery High Dose (Active Comparator): High-Dose Group: 0.4 mg/mL temsirolimus (including 20% contrast) Patients qualifying for enrollment will be randomized 2:1 for inclusion in either the treatment (low-dose or high-dose) or the control group. The first 20 patients randomized to treatment will receive low-dose. After the first 30 patients (20 low-dose and 10 control) are enrolled in the trial, enrollment will be held until 30-day safety endpoints are met, at which point the dosage will be escalated to the high dose and the trial will resume, with the remaining 30 patients randomized 2:1 for high-dose or control.
  Interventions: Drug: Temsirolimus
- Active Comparator: Temsirolimus Delivery Low Dose (Active Comparator): Low-Dose Group: 0.1 mg/mL temsirolimus (including 20% contrast) Patients qualifying for enrollment will be randomized 2:1 for inclusion in either the treatment (low-dose or high-dose) or the control group. The first 20 patients randomized to treatment will receive low-dose. After the first 30 patients (20 low-dose and 10 control) are enrolled in the trial, enrollment will be held until 30-day safety endpoints are met, at which point the dosage will be escalated to the high dose and the trial will resume, with the remaining 30 patients randomized 2:1 for high-dose or control.
  Interventions: Drug: Temsirolimus
- Placebo Comparator: Saline Delivery (Placebo Comparator): Control Group: Saline/contrast (80% normal saline for injection:20% non-ionic contrast) The first 20 patients randomized to treatment will receive low-dose. After the first 30 patients (20 low-dose and 10 control) are enrolled in the trial, enrollment will be held until 30-day safety endpoints are met, at which point the dosage will be escalated to the high dose and the trial will resume, with the remaining 30 patients randomized 2:1 for high-dose or control.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Temsirolimus — After completion of revascularization therapy and any decision to place stents, patients will be qualified for final enrollment in the study and will be treated with the investigational drug or saline. Investigators will be blinded to assignment.
  Other Names: Torisel
  Arms: Active Comparator: Temsirolimus Delivery High Dose; Active Comparator: Temsirolimus Delivery Low Dose
Drug: Saline — After completion of revascularization therapy and any decision to place stents, patients will be qualified for final enrollment in the study and will be treated with the investigational drug or saline. Investigators will be blinded to assignment.
  Arms: Placebo Comparator: Saline Delivery

SUMMARY:
This is a prospective, multi-center, randomized, dose escalation study to document the effects of adventitial delivery of temsirolimus (Torisel) after revascularization of lesions below the knee in symptomatic patients with critical limb ischemia (CLI).

DETAILED DESCRIPTION:
This is a prospective, multi-center, randomized, dose escalation study to document the effects of adventitial delivery of temsirolimus (Torisel) after revascularization of lesions below the knee in symptomatic patients with critical limb ischemia (CLI). Up to 60 patients (20 low-dose, 20 high-dose and 20 control) at up to 15 sites in the United States. This study will assess the safety and effectiveness of Bullfrog Micro-Infusion Device adventitial deposition of temsirolimus in reducing intimal hyperplasia, inflammatory markers and composite safety endpoints in patients with clinical evidence of chronic critical limb ischemia after revascularization of one or more angiographically significant lesion(s) in below-knee popliteal or tibial vessels.

ELIGIBILITY:
Inclusion Criteria:

Screening Criteria:

* Age ≥18 years and <90 years
* Patient has been informed of the nature of the study, agrees to participate and has signed an IRB approved consent form
* Female patients of childbearing potential have a negative pregnancy test ≤7 days before the procedure and are willing to use a highly effective method of birth control (See Section 12.2) one month preceding and 12 months following study treatment
* Patient has documented chronic Critical Limb Ischemia (CLI) in the target limb from the distal segment (P3) of the popliteal artery to the ankle joint prior to the study procedure with Rutherford Category 3, 4 or 5
* Life expectancy >1 year in the Investigator's opinion

Angiographic Criteria:

* Target vessel(s) diameter ≥2 mm and ≤8 mm
* Single or multiple atherosclerotic lesion(s) ≥70% in at least one below-knee popliteal or tibial target vessel including the tibioperoneal trunk that totals up to no greater than 30 cm in length (with no greater than 5 cm length of contiguous intervening normal artery), with possible extension into the popliteal artery distal to the center of the knee joint space (the P3 segment)
* Successful revascularization of the TL with less than 30% residual stenosis, run-off down to the foot and direct in-line flow to any foot wound, if a wound is present at baseline

Exclusion Criteria:

• Screening Criteria

* Patient is already enrolled in another clinical study of systemic drug therapy or another device study that has not completed its primary endpoint
* Patient unwilling or unlikely to comply with visit schedule
* Patients who are incapable of providing consent and/or incapable of understanding the nature, significance and implications of the clinical trial
* Patient is already receiving or planned to receive systemic immunotherapy, chemotherapy, or steroids (however, inhaled steroids for asthma treatment or topical steroid uses are allowed)
* Patient has a bilirubin level of >1.5xULN
* Recent (<30 days prior to study procedure) myocardial infarction
* Cerebrovascular accident <60 days prior to the study procedure
* Planned major (above the ankle) target limb amputation
* Active foot infection; however, osteomyelitis in the toes or mild cellulitis around the perimeter of gangrene or small ulcers (<25mm) are not exclusions, but osteomyelitis of the metatarsal or more proximal region would be exclusionary
* Inability to receive temsirolimus or iodinated contrast medium due to labeled contra-indications or known sensitivity reactions Estimated glomerular filtration rate (eGFR, calculated from serum creatinine using an isotope dilution mass spectrometry (IDMS)-traceable equation) less than 30 mL/min, except for patients with end stage renal disease on chronic hemodialysis
* Stage 3 (per SVS WIfI classification) or worse heel ulcers or heel ulcers that are determined to be primarily neuropathic in nature or non-ischemic in origin

Angiographic/Procedural Criteria

* Hemodynamically significant inflow lesion (≥50% DS) or occlusion in the ipsilateral iliac, SFA, or popliteal arteries (P1 and P2) in which there is failure to successfully treat and obtain a <30% residual stenosis post-revascularization, with bailout stenting as needed (in-flow lesions should be treated prior to treating the target lesion)
* Target lesion length is >30 cm as measured from proximal normal vessel to distal normal vessel
* Total length of lesions treated during the case (including target lesion, inflow lesions, and other non-target lesions) >30 cm
* Use of alternative therapy, e.g. radiation therapy, drug-eluting stents (DES) or drug-eluting balloon/drug-coated balloons (DEB/DCB) as part of the target lesion treatment or during the previous 2 months within the target lesion
* Previously implanted stent in the TL(s)
* Aneurysm in the target vessel
* Acute thrombus in the target limb
* Failure to cross the TL with a guide wire; however, subintimal wire crossing is allowed
* Heavy eccentric or concentric calcification at target lesion, which in the judgment of the investigator would prevent penetration of the Micro-Infusion Device needle through the vessel wall

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-03-03 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Freedom from MALE-POD | Up to 30 days post-procedure
  Freedome from MALE-POD at 30 days.
Transverse-view vessel area loss percentage (TVAL%) of the target lesion | Within 6 months post-procedure
  Transverse-view vessel area loss percentage (TVAL%) of the target lesion at 6 months by quantitative vascular angiography (QVA) or prior to any TLR of the target lesion before 6 months.

SECONDARY OUTCOMES:
Freedom from a composite of all-cause death, MALE and unplanned minor amputation in target limb | Up to 30 days post-procedure
  Freedom from a composite of all-cause death within 30 days from the index procedure, major adverse limb event (MALE) of the target limb, unplanned minor amputation in the target limb, and clinically driven target lesion revascularization (CD-TLR) within 6 months.
Freedom from a composite of death, unplanned minor amputation, clinically driven TLR, and major adverse limb events (MALE) | Up to 12 months post-procedure
  Freedom from a composite of death, unplanned minor amputation, clinically driven TLR, and major adverse limb events (MALE) up to 12 months from the procedure for all subjects.
Freedom from Serious Adverse Events (SAEs) | Up to 12 months post-procedure
  Freedom from serious adverse events (SAE) to 12 months from the procedure for all subjects.
Event-free survival | Up to 12 months post-procedure
  Event-free survival to 12 months from the procedure for all subjects.
Improvement in % diameter stenosis and maximum late lumen loss (LLL) of the target lesion | Up to 6 months post-procedure
  6-month improvement % diameter stenosis (%DS) of the target lesion (TL) and the maximum late lumen loss for the lesion (LLL) will be assessed by Quantitative Vascular Angiography.
Improvement in luminal volume by intravascular ultrasound (IVUS) | Up to 6 months post-procedure
  6-month improvement in luminal volume as measured by intravascular ultrasound (IVUS) within the TL (subgroup analysis).
Composite of major amputation, target vessel occlusion or CD-TLR | Up to 12 months post-procedure
  A composite at 12 months of freedom from major amputation, target vessel occlusion, or CD-TLR.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - St. Joseph Hospital of Orange Heart and Vascular Center, Orange, California
  - Denver Veterans Administration Hospital, Denver, Colorado
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - University Hospital, Cleveland, Ohio
  - Einstein Medical Center, Philadelphia, Pennsylvania
  - Sanford Research, Sioux Falls, South Dakota
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes